CLINICAL TRIAL: NCT01219400
Title: Study of the Effect of Vildagliptin on Glucagon Counterregulation Response During Hypoglycemia in Insulin-treated Patients With Type 2 Diabetes
Brief Title: Vildagliptin and the Glucagon Response to Hypoglycemia in Insulin-Treated Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 103
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes
Keywords: DPP-4; GLP-1; Glucagon; Catecholamines; Counterregulation; Insulin-treatment; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vildagliptin (Experimental): Vildagliptin (50 mg BID) given for four weeks
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin (50 mg BID) given for four weeks
  Other Names: Galvus; 274901-16-5

SUMMARY:
The purpose of this study is to explore whether the novel therapy of type 2 diabetes, vildagliptin, which inhibits dipeptidyl peptidase-4 (DPP-4), affects glucagon counterregulation during hypoglycemia in insulin-treated patients with type 2 diabetes. Vildagliptin is given, together with the on-going insulin therapy, for one month, whereafter hypoglycemia is induced under standardized conditions, and the glucagon response is determined, and compared to that after a month of placebo treatment.

DETAILED DESCRIPTION:
Vildagliptin is an inhibitor of dipeptidyl peptidase-4 (DPP-4) and inhibits glucagon secretion and stimulates insulin secretion. This improves glycemia in subjects with type 2 diabetes with a very low risk for hypoglycemia. If hypoglycemia nevertheless develops, it is important that vildagliptin under such conditions does not inhibit glucagon secretion, since that would aggravate the hypoglycemia. It was indeed previously demonstrated in type 2 diabetes that vildagliptin dos not inhibit glucagon secretion during hypoglycemia. This study explores whether vildagliptin affects glucagon counterregulation during hypoglycemia in insulin-treated patients of type 2 diabetes. Vildagliptin is given, together with the on-going insulin therapy, for one month, whereafter hypoglycemia is induced under standardized conditions, and the glucagon response is determined, and compared to that after a month of placebo treatment. The hypoglycemia is induced bvy a standardized clamp procedure.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Insulin treatment
* Age >18 years
* HbA1c <=8.5%

Exclusion Criteria:

* Pregnancy
* Lactation
* Acute infection
* Liver disease
* Treatment with cortisol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Glucagon response to hypoglycemia | 45 min
  Change in glucagon from before hypoglycemia clamp until after 45 min

SECONDARY OUTCOMES:
Catecholamine response to hypoglycemia | 45 min
  Change in catecholamines from before hypoglycemic clamp to 45 min

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahrén, MD, PhD, Study Chair — Lund University
Locations (1):
- Lund University, Lund, Sweden